CLINICAL TRIAL: NCT01313065
Title: A Dose-Escalation Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Intravenous Infusion of VX15/2503 in Adult Patients With Advanced Solid Tumors
Brief Title: Evaluation of Safety, Tolerability, PK & PD of Intravenous VX15/2503 in Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vaccinex Inc. (Industry)
Collaborators: PPD Development, LP (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VX15/2503-01 v.9
Record Dates: First submitted 2011-03-04; First posted 2011-03-11 (Estimated); Last update posted 2014-08-13 (Estimated); Status verified 2014-08

CONDITIONS: Solid Tumors
Keywords: VX15/2503; Semaphorin 4D; SEMA4D; CD100; safety; tolerability; pharmacokinetics; pharmacodynamics; advanced solid tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- VX15/2503 (Experimental): VX15/2503 monoclonal antibody at a concentration of 0.3 mg/kg - 20 mg/kg to be administered intravenously on a weekly dosing cycle.
  Interventions: Drug: VX15/2503

INTERVENTIONS:
Drug: VX15/2503 — Dose escalation will begin at low doses and will gradually increase in each future cohort. The current trial design provides for 7 study cohorts with a 20 mg/kg expansion phase.

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of IV administration of VX15/2503 in patients with advanced solid tumors. The escalation part of the study will determine the maximum tolerated dose (MTD).

DETAILED DESCRIPTION:
VX15/2503-01 is a dose-escalation, open label study to evaluate the safety and tolerability of IV administered VX15/2503 in patients with advanced solid tumors. This will be accomplished by using a dose escalation procedure starting at low doses of VX15/2503 and will continue based on predefined parameters until the maximum tolerated dose is identified.

The study drug, VX15/2503, is a monoclonal antibody that binds to the semaphorin 4D (SEMA4D; CD100) antigen. Semaphorins have been shown to play an important role in certain physiological processes such as vascular growth, tumor progression and immune cell regulation. Experimental evidence suggests that SEMA4D has two mechanisms of action that result in angiogenesis and tumor proliferation and invasion. Antibody neutralization of SEMA4D thus may represent a new therapeutic strategy for cancer treatment.

ELIGIBILITY:
Main Inclusion Criteria:

* Patients 18 yrs or older with confirmed histological or cytological advanced solid tumors, relapsed or refractory to standard treatment for which no curative therapy is available; patients must demonstrate progressive disease prior to entry
* Has measurable disease as defined by RECIST1.1
* Life expectancy of at least 3 months (per investigator assessment)
* ECOG performance status of 0-2
* Adequate bone marrow, renal and liver function
* Recovered from any significant prior toxicity of previous anti-neoplastic therapy
* For patients of reproductive potential, is willing to use a medically acceptable form of contraception throughout the study period and for at least 4 weeks after the last dose of VX15/2503
* Expansion cohort - patients in this cohort must have one of the following characteristics:
* A diagnosis of a pancreatic neuroendocrine tumor OR
* A diagnosis of a soft tissue sarcoma OR
* A diagnosis of a bone metastasis OR
* A diagnosis of advanced solid tumor AND a T cell count of at least 1500 cells/uL OR a B cell count of at least 250 cells/uL at screening

Main Exclusion Criteria:

* Treatment with anti-neoplastic agents (chemotherapy, immunotherapy, radiotherapy or endocrine therapy) within 3 weeks prior to start of study treatment
* Treatment with an investigational agent within 4 weeks prior to start of study treatment
* Is on concurrent anti-neoplastic therapy with the exception of continuing luteinizing hormone-releasing hormone agonist/antagonist therapy for patients with castrate-resistant prostate cancer
* Treatment with oral or parenteral corticosteroids in excess of 10mg/day of prednisolone or equivalent for more than 5 days within 4 weeks prior to start of study treatment or a requirement for systemic immunosuppressive therapy for any reason
* Untreated brain Mets or CNS tumor involvement
* Any other intercurrent illness or condition which could impact patient compliance or ability to complete the study
* Sensitivity to VX15/2503 or the ingredients or excipients of VX15/2503
* Pregnant or breast-feeding women (women of child-bearing potential must have negative serum pregnancy test within 3 days prior to receiving the first dose of VX15/2503)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2011-01; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Safety/tolerability as measured by number of patients with adverse events | Up to 18 months
  Subject incidence of treatment-emergent adverse events
Maximum tolerated dose as measured by frequency of dose limiting toxicities | Four (4) weeks after first dose

SECONDARY OUTCOMES:
Peak plasma concentration (Cmax) of VX15/2503 | Four (4) hours after start of infusion
Area under the plasma concentration versus time curve (AUC) of VX15/2503 | Up to seven (7) days after first dose
Half-life of VX15/2503 | Up to 14 days after first dose

OTHER OUTCOMES:
SEMA4D T cell percent saturation of VX15/2503 | Up to 18 months
Number of patients who develop anti-drug antibody | Up to 18 months
Overall response rate (ORR) using RECIST 1.1 | Up to 18 months
Progression-free survival (PFS) using RECIST 1.1 | Up to 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Amita Patnaik, MD, Principal Investigator — South Texas Accelerated Research Therapeutics, LLC; Ramesh K Ramanathan, MD, Principal Investigator — TGen Clinical Research Service at Scottsdale Healthcare
Locations (2):
- United States (2):
  - Virginia G. Piper Cancer Center at Scottsdale Healthcare, Scottsdale, Arizona
  - South Texas Accelerated Research Therapeutics, LLC, San Antonio, Texas

REFERENCES:
- [Derived] Worzfeld T, Offermanns S. Semaphorins and plexins as therapeutic targets. Nat Rev Drug Discov. 2014 Aug;13(8):603-21. doi: 10.1038/nrd4337. PMID 25082288